CLINICAL TRIAL: NCT03988556
Title: Feasibility and Safety of CareMin650 in Cancer Patients at High Risk of or Suffering From Oral Mucositis and/or Radiation Dermatitis Due to the Administration of Radiotherapy: A Prospective Non-comparative Study
Brief Title: Feasibility and Safety of CareMin650 in Patients at Risk of or Suffering From Oral Mucositis and/or Radiation Dermatitis
Acronym: SafePBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoMedLight (Industry)
Collaborators: Qualissima (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID-RCB: 2018-A03356-49
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Oral Mucositis Due to Radiation; Radiation Dermatitis
Keywords: Photobiomodulation; Oral Mucositis; Radiation Dermatitis; Radiotherapy; Head and neck cancer; Breast cancer
MeSH Terms: conditions — Radiodermatitis; Stomatitis; Head and Neck Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A1 - Head & neck cancer - Prophylactic intent (Experimental): Patients with head & neck cancer starting radiotherapy +/- chemotherapy +/- targeted therapy (no lesions, prophylactic intent).
  Treatment with CareMin650 will start on the first day of radiotherapy and will be administered during the whole radiotherapy period (6 to 8 weeks maximum), ideally 5 days/week, at least 3 days/week, before or after the radiotherapy session.
  The device will be used on irradiated areas presenting a risk of radiotherapy-related complications. The prophylactic treatment will aim at preventing both oral mucositis and radiodermatitis.
  .
  Interventions: Device: Photobiomodulation using CareMin650 at 3 Joules (prophylactic intent)
- Cohort A2 - Head & neck cancer - Curative intent (Experimental): Patients with head & neck cancer having started radiation therapy and presenting with grade 1 to 3 lesions of oral mucositis and/or radiation dermatitis (curative intent).
  Treatment with CareMin650 will start as soon as the lesion is diagnosed and will be administered at each radiotherapy session, during the whole radiotherapy period (6 to 8 weeks maximum).
  The device will be used on each lesion. All existing lesions will be treated whether they are oral mucositis or radiodermatitis lesions.
  Interventions: Device: Photobiomodulation using CareMin650 at 6 Joules (curative intent)
- Cohort B1 - Breast cancer - Prophylactic intent (Experimental): Patients with breast cancer starting radiation therapy (i.e. no lesions, prophylactic intent).
  Treatment with CareMin650 will start on the first day of radiotherapy and will be administered during the whole radiotherapy period (6 to 8 weeks maximum), ideally 5 days/week, at least 3 days/week, before or after the radiotherapy session.
  The device will be used on irradiated areas presenting a risk of radiotherapy-related complications. The prophylactic treatment will aim at preventing radiodermatitis.
  Interventions: Device: Photobiomodulation using CareMin650 at 3 Joules (prophylactic intent)
- Cohort B2 - Breast cancer - Curative intent (Experimental): Patients with breast cancer having started radiation therapy and presenting with grade 1 to 3 lesions of radiation dermatitis (curative intent).
  Treatment with CareMin650 will start as soon as the lesion is diagnosed and will be administered at each radiotherapy session, during the whole radiotherapy period (6 to 8 weeks maximum).
  The device will be used on each lesion. All existing lesions will be treated.
  Interventions: Device: Photobiomodulation using CareMin650 at 6 Joules (curative intent)

INTERVENTIONS:
Device: Photobiomodulation using CareMin650 at 6 Joules (curative intent) — CareMin650 is a photobiomodulation device which consists of a Lightbox and a light applicator to deliver red light with wavelength of 650 nm and irradiance between 10 and 50 mW/cm² to skin or mucosa.
  For curative treatment, the dose to be delivered has been set at 6J/cm2. If the lesions of patients included in a curative cohort are resolved before the end of the radiotherapy period, the treatment will be applied with a preventive aim and the dose will decrease from 6 to 3J/cm2.
  Arms: Cohort A2 - Head & neck cancer - Curative intent; Cohort B2 - Breast cancer - Curative intent
Device: Photobiomodulation using CareMin650 at 3 Joules (prophylactic intent) — CareMin650 is a photobiomodulation device which consists of a Lightbox and a light applicator to deliver red light with wavelength of 650 nm and irradiance between 10 and 50 mW/cm² to skin or mucosa.
  For prophylactic treatment, the dose to be delivered has been set at 3J/cm2. If oral mucositis or radiodermatitis occurs in a patient included in a prophylactic cohort, the lesions will be treated with a curative intent and the dose will increase from 3 to 6J/cm2.
  Arms: Cohort A1 - Head & neck cancer - Prophylactic intent; Cohort B1 - Breast cancer - Prophylactic intent

SUMMARY:
The main objective of the present study is to investigate the feasibility, safety and tolerability of CareMin650 in patients with 1) head & neck cancer at high risk of or suffering from oral mucositis and/or radiation dermatitis due to the administration of radiotherapy with or without chemotherapy with or without targeted therapy, 2) breast cancer at high risk of or suffering from radiation dermatitis due to the administration of radiotherapy.

DETAILED DESCRIPTION:
The main objective of the present study is to investigate the feasibility, safety and tolerability of CareMin650 in patients with 1) head & neck cancer at high risk of or suffering from oral mucositis and/or radiation dermatitis due to the administration of radiotherapy with or without chemotherapy with or without targeted therapy, 2) breast cancer at high risk of or suffering from radiation dermatitis due to the administration of radiotherapy.

This is a prospective non-comparative study. Two cohorts of patients will be included, based on the tumour location. Each cohort will be divided into two subgroups according to whether the treatment is for curative or preventive purposes.

* Patients with head & neck cancer (cohort A), either starting radiotherapy with or without chemotherapy with or without targeted therapy (no lesions, prophylactic intent, cohort A1) or having started treatment and presenting with grade 1 to 3 lesions of oral mucositis and/or radiation dermatitis (curative intent, cohort A2).
* Patients with breast cancer requiring radiation therapy (cohort B), either starting radiation therapy (i.e. no lesions, prophylactic intent, cohort B1) or having started treatment and presenting with grade 1 to 3 lesions of radiation dermatitis (curative intent, cohort B2) it is planned to select a maximum number of 72 patients (36 in each cohort)

Consecutive patients will be included in each of the four predefined subgroups, until the target number of patients in each subgroup has been reached.

The photobiomodulation treatment will be initiated at inclusion and will be continued for the duration of radiotherapy (6 to 8 weeks maximum).

The maximum total participation in the study is anticipated to be approximately ten weeks for each patient.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria common to both cohorts:

* Adult patients (age ≥18 years) accepting to participate in the study and having signed the written informed consent form prior to any protocol-specific procedures.
* Having an ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2.
* Having a life expectancy greater than 3 months according to the investigator medical judgement.
* Having the ability to understand and sign the written informed consent form and willing to comply with protocol requirements.

Specific criteria for inclusion in head and neck cancer cohort (cohort A):

* Patient with histologically proven squamous cell carcinoma of oropharynx, nasopharynx, hypopharynx, larynx or oral cavity with or without prior surgical resection
* Patient with dental examination prior to chemo-radiotherapy and any required dental treatment performed
* In cohort A1 (patient with no oral mucosa or skin lesion, starting radiotherapy), patient scheduled to receive intensity modulated radiation therapy on at least 50% of the oral mucosa at a total dose of at least 40 Gy, alone or associated with chemotherapy or targeted therapies.
* In cohort A2, (on-going radiotherapy), presence of oral mucositis and/or radiation dermatitis grade 1, 2 or 3.

Specific criteria for inclusion in breast cancer cohort (cohort B)

* Patient with histologically proven breast cancer
* After breast-conserving surgery, or total mastectomy if the patient is at high risk of radiodermatitis based on the investigator's judgement.
* In cohort B1, (patient with no skin lesion starting radiotherapy) patient scheduled to receive radiation therapy.
* In cohort B2 (on-going radiotherapy) presence of radiation dermatitis grade 1, 2 or 3.

Exclusion Criteria:

Exclusion Criteria common to both cohorts:

* Any condition that may interfere with adherence to treatment according to the investigator's judgment
* Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.
* Patient with a known polyurethane allergy
* Females patients who are pregnant or breastfeeding
* Female patients who do not fall into 1 of the following categories:

  * Post-menopausal
  * Surgically sterile
  * Using one of the following birth control methods throughout the duration of the study:

    * Intrauterine device (> 14 days)
    * Barrier method (condom or diaphragm) with spermicide (> 14 days)
    * Hormonal contraception (same dose and same formulation for at least 6 months)
* Patient participating in another clinical trial involving drugs or non-drug therapies aiming to treat or prevent lesions induced by radiotherapy

Specific criteria for non inclusion in head and neck cancer cohort (coh ort A):

* Active bleeding, coagulopathy or pathologic condition that would confer a high risk of bleeding
* Hb < 8g/dL; neutrophils < 1000 mm3; platelets < 50 000/mm3

Specific criteria for non inclusion in breast cancer cohort (cohort B):

* Previous irradiation to the same breast
* Any pre-existing skin disorders located on the chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Occurence of adverse events | Continuous (from screening visit to Follow-up visit (10 weeks maximum) + 30 days )
  This safety outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatments.
Rate of discontinuation due to AEs | Continuous on 6 to 8 weeks maximum (Inclusion visit to End of radiotherapy visit)
  Rate of discontinuation due to AEs.

SECONDARY OUTCOMES:
Skin lesions assessment - time of lesion occurrence | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  time of lesion occurrence
Skin lesions assessment - size of lesions | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  size of lesions (centimeters square)
Skin lesions assessment - location | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  location
Skin lesions assessment - Grade | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Severity grade according to CTCAE V3 (0 (absence) to 5 (death))
Skin lesions assessment - Time until resolution | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Time until resolution (defined as lesions that do not require further treatment).
Oral mucosa lesions assessment - time of lesion occurrence | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  time of lesion occurrence
Oral mucosa lesions assessment - size of lesions | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  size of lesions (centimeters square)
Oral mucosa lesions assessment - location | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Location
Oral mucosa lesions assessment - Grade | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Severity grade according to CTCAE V3 (0 (absence) to 5 (death))
Oral mucosa lesions assessment - Time until resolution | Inclusion visit, before each therapeutic session with the device (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Time until resolution (defined as lesions that do not require further treatment).

OTHER OUTCOMES:
Score at visual analogic scale of pain | Inclusion visit, first therapeutic session with the device of each radiotherapy week (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  score at visual analogic scale of pain (continuous values from 0 to 10) completed by patients
Analgesic consumption | Inclusion visit, first therapeutic session with the device of each radiotherapy week (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Assessment of patients analgesic consumption for the pain induced by the oral mucositis and/or radiation dermatitis lesion(s)
Xerostomia assessment | First therapeutic session with the device of each radiotherapy week (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Assessment of xerostomia grade (0 to 3)
Food intake | Inclusion visit, first therapeutic session with the device of each radiotherapy week (6 to 8 weeks maximum), end of radiotherapy visit (after 6 to 8 weeks maximum), Follow-up visit (7 to 13 days after last exposition)
  Assessment of oral lesion(s) consequences on food intake
Patients quality of life | 2 times: Inclusion visit, end of radiotherapy visit (after 6 to 8 weeks maximum)
  SF-12 questionnaire score (12 questions, 2 subscores: mental quality of life score and physical quality of life score) assessed by patients
Patients satisfaction | 1 time: end of radiotherapy visit (after 6 to 8 weeks maximum)
  Questionnaire of satisfaction (developed by the sponsor; 9 questions on pain, comfort, duration of sessions, ability to hold the device alone and global satisfaction) completed by patients
Convenience of the device and satisfaction of the operator | 1 time: end of radiotherapy visit (after 6 to 8 weeks maximum)
  questionnaire of convenience of the device and satisfaction (developed by the sponsor; 12 questions on use, experience with the device, technical settings, duration of sessions and global recommendations) completed by health professionals
ECOG Scale of Performance Status | 2 times: Inclusion visit, end of radiotherapy visit (after 6 to 8 weeks maximum)
  ECOG (Eastern Cooperative Oncology Group) performance status (score from 0 to 5) assessed by the investigator
Use of the device - Number of sessions | throughout the entire treatment period with the device (Day 1 until 6 to 8 weeks maximum)
  Number of therapeutic sessions with the device
Use of the device - Frequency of use | throughout the entire treatment period with the device (Day 1 until 6 to 8 weeks maximum)
  Frequency of therapeutic sessions with the device
Use of the device - Cumulative duration of use | throughout the entire treatment period with the device (Day 1 until 6 to 8 weeks maximum)
  Cumulative duration of procedures
Use of the device - Cumulative dose | throughout the entire treatment period with the device (Day 1 until 6 to 8 weeks maximum)
  Cumulative dose delivered

CONTACTS AND LOCATIONS:
Overall Officials: René-Jean Bensadoun, MD, Principal Investigator — Centre de Haute Energie - Nice
Locations (5):
- France (5):
  - Institut de radiothérapie et radiochirurgie Hartmann, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Centre de Haute Energie, Nice
  - Institut Curie, Paris
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of Neomedlight — http://www.neomedlight.com/